CLINICAL TRIAL: NCT04817631
Title: Management of Tuba-ovarian Abscess: a 10 Year Single-center Experience
Brief Title: Management of Tubo-ovarian Abscess: a Single Center Experience
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Nura Fitnat Topbas Selcuki, MD, Specialist in Obstetrics and Gynecology, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: TOA
Record Dates: First submitted 2021-03-14; First posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Tubo-ovarian Abscess
Keywords: abscess drainage; abscess size; medical treatment; surgical treatment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: tuboovarian abscess — Evaluating the surgical and medical management of tuboovarian abscess

SUMMARY:
Electronic database of our tertiary obstetrics and gynecology clinic was searched for patients who were treated for tub-ovarian abscess during the last 10 years (January 2010- November 2020). Patients' biometric data, admission date and duration, medical and surgical treatment modalities were recorded using an Excel sheet. Patients will be evaluated on the basis of the treatment they receive, length of treatment, if surgically treatment the type of surgery performed. Hospitalization length, readmission, recurrence will be compared between treatment modalities.

DETAILED DESCRIPTION:
This retrospective study is conducted at Health Sciences University Turkey, Sisli Hamidiye Etfal Training and Research Hospital Department of Obstetrics and Gynecology. Electronic database was searched for patients who were treated for tub-ovarian abscess during the last 10 years (January 2010- November 2020). Patients' biometric data, admission date and duration, medical and surgical treatment modalities were recorded using an Excel sheet. Patients will be evaluated on the basis of the treatment they receive, length of treatment, if surgically treatment the type of surgery performed. Hospitalization length, readmission, recurrence will be compared between treatment modalities. A change in management strategy over the years if any will be reported.

ELIGIBILITY:
Inclusion Criteria:

* presence of a pelvic mass > 3 cm with transvaginal ultrasound or magnetic resonance imaging indication abscess
* cervical and uterine tenderness
* abdominal rebound-defense under physical examination indication peritoneal irritation
* presence of symptoms such as fever, pelvic pain and increase in laboratory infection parameters

Exclusion Criteria:

* Patients with known malignities
* Patients with incomplete data in the clinic's electronic database
* Patients who continued their treatment at other centers

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — the study will be conducted on female patients with tuboovarian abscess
Study Population: Women over 18 years of age who presented to our clinic with symptoms of infection and where tuboovarian abscess was suspected with physical and ultrasonographic examination are included in this study
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Evaluating the management of tuboovarian abscess on the basis of surgical or medical modalities by assessing hospitalization duration and recurrence | 10 years
  Patients' demographics data (age, gravity, parity, presence of additional comorbidities and BMI) will be recorded. Their laboratory assessment of infection prior to treatment begin such as CRP an procalcitonin will be recorded. Their treatment modalities in terms of surgery or antibiothepry, duration of hospitalization and recurrence will be recorded. Statistical analysis will be done using SPSS. Student's t test will be used for comparison where necessary. Significance will be evaluated using p-value.

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No